CLINICAL TRIAL: NCT03998111
Title: The Role of Genetic Variation in CLTCL1 and Other Related Genes in Relation to Whole-body Glucose Control: A Pilot Study
Brief Title: Genetic Variation in CLTCL1 and Whole-body Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier Gonzalez (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor-Investigator, Javier Gonzalez, Senior Lecturer, University of Bath
Organization: University of Bath (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EP 17/18 252
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Glucose Control
Keywords: Glucose; Genetic variation; CHC22; CLTCL1
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial (Experimental): Participants will undergo one trial visit where they will ingest an oral glucose load diluted in solution (oral glucose tolerance test) and blood samples will be measured over the following 2-hours. The buffy coat layer from the baseline sample will be obtained to extract DNA.
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — Participants will ingest 75 g anhydrous glucose dissolved in water and the blood responses will be measured over the following 2-hours using a venous cannula.

SUMMARY:
Maintaining stable blood glucose concentrations after eating has important implications for health. Individuals who are better able to maintain stable blood glucose concentrations after consuming carbohydrate have a lower risk of mortality from cardiovascular disease. Muscle is the primary tissue for glucose disposal following a meal, and responsiveness of this tissue to insulin is dictated by GLUT4 translocation to the muscle cell membrane. Clathrin heavy chain isoform 22 (CHC22) is a protein that plays a key role in intracellular GLUT4 action, and it may play an important role in whole-body glucose control. Genetic variation in the gene which codes for CHC22 may be able to explain differences in glucose control at the whole-body level.

DETAILED DESCRIPTION:
The ability to maintain relatively stable blood glucose concentrations after eating has important implications for health. Individuals who are better able to maintain stable blood glucose concentrations after consuming carbohydrate have a lower risk of mortality and morbidity from cardiovascular disease. Muscle is the primary tissue for glucose disposal after a meal and the ability to tolerate a glucose load is largely dependent on the ability of muscle to respond to insulin by translocating the glucose transporter, GLUT4, to the muscle cell membrane, facilitating glucose import into muscle from the circulation. Therefore, by understanding the mechanisms that explain why some people are better able to maintain glucose control can give insight into how to target physiological pathways (such as muscle glucose uptake) to reduce disease risk and improve health.

Clathrins are cytoplasmic proteins that play essential roles in cell membrane trafficking pathways. Pilot data indicate that the clathrin heavy chain isoform 22 (CHC22) plays a key role in intracellular targeting of GLUT4 and may therefore play an important role in whole-body glucose control. Cell-based studies suggest that genetic variation in the CLTCL1 gene (which encodes for CHC22) at SNP rs1061325, influences GLUT4 retention. It is currently unknown whether genetic variation in CHC22 has consequences for whole-body glucose control in humans.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.5-29.9 kg/m^2
* Aged 18-65 years
* Able and willing to provide informed consent and safely comply with study procedures

Exclusion Criteria:

* Any reported condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias
* Any diagnosed metabolic disease (e.g. type 1 or type 2 diabetes)
* Any reported use of substances which may pose undue personal risk to the participants or introduce bias into the experiment
* Lifestyle not conforming to standard sleep-wake cycle (e.g. shift worker)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Plasma glucose incremental area under the curve (CHC22 genotype) | 2 hours
  Plasma glucose samples will be obtained throughout the 2-hour postprandial period and the incremental area under the curve will be calculated, this will be grouped by CHC22 genotype.
Peak plasma glucose (CHC22 genotype) | 2 hours
  Plasma glucose samples will be obtained throughout the 2-hour postprandial period and the peak glucose concentration will be measured, this will be grouped by CHC22 genotype.

SECONDARY OUTCOMES:
Fasting plasma glucose concentrations (CHC22 genotype) | 2 hours
  Plasma glucose will be measured at baseline and will be grouped by CHC22 genotype.
Plasma glucose incremental area under the curve (other genotypes) | 2 hours
  Plasma glucose samples will be obtained throughout the 2-hour postprandial period and the incremental area under the curve will be calculated, this will be grouped by genotyping other genes related to glucose control or sweet taste sensitivity.
Fasting plasma glucose concentrations (other genotypes) | 2 hours
  Plasma glucose will be measured at baseline and will be grouped by genotypes related to glucose control and sweet taste sensitivity.
Matsuda insulin sensitivity index | 2 hours
  Matsuda insulin sensitivity index will be calculated using blood samples collected in the 2-hour postprandial period.
Homeostasis model of insulin resistance | 2 hours
  Homeostasis model of insulin resistance will be calculated using blood samples collected in the 2-hour postprandial period.

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom